CLINICAL TRIAL: NCT07310563
Title: A Phase 1, Randomized, Open-label, Parallel-group, Drug-drug Interaction Study to Evaluate the Effect of Antiemetic Medication on the Pharmacokinetics of AMG 133 in Participants Living With Overweight or Obesity
Brief Title: A Trial to Evaluate Interactions Between Antiemetic Medication and AMG 133 in Participants Living With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20210281
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity
Keywords: Antiemetic; Drug-drug Interaction; AMG 133; Ondansetron; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Ondansetron

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Dose AMG 133 without Ondansetron (Experimental): Participants will receive a single subcutaneous (SC) low dose of 70 mg AMG 133.
  Interventions: Drug: AMG 133
- High Dose AMG 133 without Ondansetron (Experimental): Participants will receive a single SC high dose of 350 mg AMG 133.
  Interventions: Drug: AMG 133
- Low Dose AMG 133 with Ondansetron (Experimental): Participants will receive a single SC low dose of 70 mg AMG 133 and ondansetron 8 mg orally disintegrating tablet (ODT) every 8 hours for 72 hours.
  Interventions: Drug: AMG 133; Drug: Ondansetron
- High Dose AMG 133 with Ondansetron (Experimental): Participants will receive a single SC high dose of 350 mg AMG 133 and ondansetron 8mg ODT every 8 hours for 72 hours.
  Interventions: Drug: AMG 133; Drug: Ondansetron

INTERVENTIONS:
Drug: AMG 133 — AMG 133 will be administered SC.
Drug: Ondansetron — Ondansetron will be administered via ODT.
  Arms: High Dose AMG 133 with Ondansetron; Low Dose AMG 133 with Ondansetron

SUMMARY:
The primary objective of this trial is to evaluate the pharmacokinetics (PK) of AMG 133 administered alone and in combination with an antiemetic medication, ondansetron, in participants living with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria

1. Male or female participants, between 18 and 65 years of age.
2. Body mass index > 25 kg/m^2.

Exclusion Criteria

1. History or evidence of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the Investigator, would pose a risk to participant safety or interfere with the trial evaluation, procedures, or completion.
2. History of or active diabetes or hemoglobin A1C > 6.5%.
3. History or evidence of endocrine disorder.
4. History of acute or chronic pancreatitis within 1 year, or elevation in serum lipase/amylase (> 2 x upper limit of normal [ULN]), or fasting serum triglyceride level of > 500 mg/dL.
5. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2.
6. Uncontrolled thyroid disease.
7. History or current signs or symptoms of cardiovascular disease.
8. A QT interval corrected for heart rate based on the Fridericia's method (QTcF) interval > 450 msec in male participants or > 470 msec in female participants or history/evidence of long QT syndrome.
9. History of hypersensitivity, intolerance, or allergy to AMG 133 or its ingredients.
10. Any contraindication to ondansetron ODT according to the applicable labelling.
11. Alanine aminotransferase or aspartate aminotransferase > 2 x the ULN.
12. Use of any over-the-counter or prescription medications within 30 days or 5 half-lives (whichever is longer) before check-in.
13. Current use or prior use of any glucagon-like peptide 1 receptor (GLP-1R) agonist, or glucose-dependent insulinotropic polypeptide receptor (GIPR) agonist or antagonist within the past 3 months.
14. Participant has received a dose of an investigational medicinal product (IMP) within the past 30 days or 5 half-lives.
15. Have previously completed or withdrawn from this trial or any other trial investigating AMG 133 or have previously received the IMP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of AMG 133 | Up to Day 120
Area Under the Plasma Concentration-time Curve (AUC) from Time Zero to Time of Last Quantifiable Concentration (AUClast) of AMG 133 | Up to Day 120
AUC from Time Zero to Infinity (AUCinf) of AMG 133 | Up to Day 120

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 120
Number of Participants with Serious AEs (SAEs) | Up to Day 120
Number of Participants with Anti-AMG 133 Antibodies | Up to Day 120

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- CenExel Collaborative Neuroscience Research, LLC Los Alamitos, Los Alamitos, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com